CLINICAL TRIAL: NCT05377008
Title: Preliminary Feasibility and Clinical Effectiveness of a Single-Session Intervention on the Neurocognitive Functioning of Children and Adolescents With Neurofibromatosis Type 1
Brief Title: Intervention Effectiveness on the Neurocognitive Functioning of Children and Adolescents With Neurofibromatosis Type 1
Acronym: OPTIMAL-SSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: HM20024159
Record Dates: First submitted 2022-05-05; First posted 2022-05-17 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Neurocognitive Deficit; Mental Health Impairment; Neurofibromatosis 1
Keywords: Neurofibromatosis; Neurocognitive; Intervention
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility study comprising a randomized controlled trial involving 50 families (i.e., parent/guardian AND child ages 6 to 16 years with NF). Consented participants will be randomly allocated to the intervention (n=25) or control (n=25) arms.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patient randomization is assigned after baseline is completed (i.e., the patient and assessor are not aware of random assignment until after the baseline is completed). The Principal Investigator and Clinical Research Coordinator will be the only ones with access to random assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Parents in the intervention arm will receive one single-session intervention one month after completion of baseline measures. They will also complete a feasibility exit interview one month after completion of their data collection period (i.e., at 7 months).
  Interventions: Behavioral: OPTIMAL-SSI
- Control (No Intervention): Families in the control arm will complete measures at the exact same timepoints as those in the intervention arm but will not receive the single session intervention and will not complete the feasibility exit interview. They will receive the same information as the intervention arm via an education manual at the completion of their data collection period.

INTERVENTIONS:
Behavioral: OPTIMAL-SSI — The purpose of the intervention feedback session will be twofold: 1) to provide the results of the previous assessment, and 2) to provide general psychoeducation on psychological and neurocognitive functioning and tailored cognitive and behavioral interventions based on the results in order to reduce the impact of psychological and neurocognitive deficits.
  Arms: Intervention

SUMMARY:
Children with neurofibromatosis are more likely to have difficulties related to their psychological and neurocognitive functioning (e.g., more likely to have depression, have social difficulties, be diagnosed with ADHD). The purpose of this randomized control study is to determine how effective and useful this study's single session intervention can be in improving psychological and neurocognitive functioning. Enrolled families will consist of one parent/guardian and child. Parents and patients will complete questionnaires and objective tests at baseline, 3 months, and 6 months. Families randomized to the intervention arm will be provided with one single session intervention at Month 1 to learn about their child's testing results and receive psychoeducation and recommendations related to psychological and neurocognitive functioning.

DETAILED DESCRIPTION:
Neurofibromatosis type 1 (NF1) is a chronic illness that is typically diagnosed during childhood and is associated with a variety of medical, psychological, and neurocognitive symptoms. NF1 is a genetic disorder, affecting about 1 in 3,000 people throughout the world. Diagnosis usually occurs in childhood and is characterized by the presence of several markers, including, but not limited to: multiple café au lait (light brown) skin spots, neurofibromas (small benign growths) on or under the skin, optic pathway gliomas, bone dysplasia, and freckling in the armpits or groin. Aside from its medical manifestations, NF1 also is associated with psychological impairment and a wide variety of neurocognitive deficits. In comparison to healthy peers and the general population, children and adolescents with NF1 have been found to have more social difficulties (e.g., more peer conflicts, fewer friends), internalizing symptoms (e.g., anxiety, depression, withdrawal), externalizing symptoms (e.g., sub-threshold or clinical symptoms consistent with ADHD such as inattention, hyperactivity, impulsivity), sleep difficulties; and worse quality of life. Additionally, while the vast majority of children with NF1 have intelligence in the average to low average range, neurocognitive deficits have been found in a range of domains including: linguistic development, verbal concept formation, reasoning, visuospatial skills, motor skills, executive function (e.g., cognitive flexibility, working memory, inhibitory control), academic achievement (e.g., reading/spelling, math), and attention. There is further support that early onset of mental health problems are associated with both future mental health problems and poorer functional outcomes in adulthood (e.g., unemployment, lower earnings, lower academic attainment).

Children with NF are more likely to be diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) than their healthy counterparts. Early detection, prevention, and intervention of psychological and neurocognitive risk may serve as a protective factor for later adverse outcomes. A meta-analysis of 175 research studies worldwide on ADHD in children ages 18 and younger found an overall pooled estimate of 7.2% of children and adolescents diagnosed with ADHD within the general population; however, ADHD is over-represented within the NF1 population, with an estimated 31 to 50% of children meeting diagnostic criteria for ADHD. Although there is limited research investigating the longitudinal impact of ADHD and NF on pediatric patients, longitudinal studies of children with ADHD document deficits in multiple domains including lower levels of education, poorer social functioning, and worse occupational outcomes. Therefore, children with comorbid diagnoses of both NF1 and ADHD or even those NF patients with sub-threshold symptoms of ADHD are likely to be at an increased risk for functional deficits later in life.

Given the general current demand for psychological services, there is a great need for brief, problem-focused psychological interventions targeting psychological and neurocognitive functioning in NF. Emerging data indicate a significant increase in mental health needs as a result of the COVID-19 pandemic, which is consistent with previous large-scale disasters and pandemics. This is a significant healthcare crisis given that prior to the pandemic in the United States, more than 11.8 million people reported having unmet mental health needs. This translates to more individuals needing mental health intervention without access; and, subsequently challenges mental health providers to expand services through novel models of intervention delivery (e.g., delivering brief problem-focused interventions based on findings from standardized assessments in unconventional settings, such as, during multidisciplinary medical visits for their medical condition). One novel delivery method of psychological services is the single-session intervention (SSI), which is defined as the intentional delivery of one visit or encounter with a clinic, provider, or program. Although there is no current research investigating the feasibility and clinical effectiveness of SSI's for pediatric patients diagnosed with NF, a meta-analysis of 50 randomized control trials of SSI's for youth with psychological problems showed a significant beneficial effect (g=0.32), with greatest effect sizes for reducing anxiety (g=0.56) and conduct problems (g=0.54). Although psychoeducation-based SSI's often were found to have a small effect size, a systematic review of 13 studies conducted between 1990 and 2018 that investigated the effects of psychoeducation-based interventions on youth with ADHD showed moderate to large effects on ADHD symptom improvement as reported by parents/teachers (g=0.787), and parent/teacher and child knowledge about ADHD (g=1.037 and g=0.721, respectively).

This is a pilot feasibility study comprising a randomized controlled trial involving patients' ages 6 to 16 years (n=50) with NF. Patients will complete standardized assessment batteries and questionnaires assessing their neurocognitive, executive, and psychological functioning. The present study will yield longitudinal patterns of neurocognitive and psychosocial outcomes across the six month period, and, collect data for preliminary development of a single session intervention. In order to gather information on how patients perform and behave in different settings, patients, parents, and teachers will also complete standardized questionnaires to gather information on psychological functioning over a six month period. Given NF is associated with psychological impairment and a wide variety of neurocognitive deficits, as well as poorer functional outcomes in adulthood, there is a great need for early detection, prevention, and intervention for this vulnerable patient population.

The proposed study has the following specific aims: Aim 1) Examine the preliminary feasibility and acceptability of using a single-session intervention focused on psychoeducation and cognitive behavioral-based recommendations related to psychological, neurocognitive, and executive functioning over six months. Hypothesis 1a: We hypothesize that families will report high acceptability for the intervention. Hypothesis 1b: It is hypothesized that families assigned to the intervention group will demonstrate improvements in both objective and subjective assessments of psychological and neurocognitive symptoms, e.g., inattention and impulsivity, as well as, executive functioning when compared to those in the control group. Aim 2) Examine descriptive and longitudinal patterns of psychological and neurocognitive factors (e.g., intellectual functioning, executive functioning, attention) across six months for the sample overall, as well as, for those in the intervention and control groups. Hypothesis 2a: It is hypothesized that a similar prevalence of ADHD for patients with NF that is seen in the literature (i.e., between 31-50%) will also be observed in our sample. Hypothesis 2b: It is hypothesized that there will be individual differences in neurocognitive patterns (e.g., executive functioning, attention) across six months in pediatric patients with neurofibromatosis (NF) with significant intra-sample variability, including differences observed between those who participated in the intervention versus those who did not. We suspect that there will be subgroups of patients who have increases in attention difficulties and executive function deficits over time, another subgroup will have decreases in attention difficulties and executive function deficits over time, and a subgroup who will have stable patterns across six months.

STUDY DESIGN

Approach:

Overview of Study Design: The current design is a pilot feasibility study comprising a randomized controlled trial involving patients ages 6 to 16 years (n=50) who are diagnosed with NF and followed by the comprehensive multidisciplinary NF clinic (Dr. Wang, Director; Dr. Rohan, Co-Director). The proposed study will contribute to new knowledge by describing trajectories of neurocognitive factors over time; as well as, examining the preliminary feasibility and effectiveness of a single-session intervention on improving psychological and neurocognitive factors such as attention and executive functioning.

This comprehensive measurement approach provides a powerful tool to address important scientific and clinically relevant questions: 1) What are the patterns of neurocognitive symptom presentation in pediatric NF?; and, how do these symptoms relate to psychosocial and health outcomes over time?; 2) How might patients and families benefit from receiving psychoeducation about neurocognitive, executive, and psychological functioning in patients with NF; as well as receiving tailored recommendations based on results of neurocognitive assessments? The use of multiple measures of neurocognitive functioning (multiple reporters and objective and subjective assessment methods), standardized questionnaires, and a single-session intervention in a pilot feasibility study of patients' ages 6 to 16 years is an innovative approach that has potential clinical utility and impact. For example, identification of neurocognitive and executive functioning deficits from multiple informants may allow development of more precise interventions in different settings for children (e.g., school, home). This approach also affords the opportunity to identify risk and protective factors in living with a chronic illness and to develop preventative and therapeutic interventions that can be delivered at the point of care to minimize barriers and maximize facilitators associated across the illness trajectory for this vulnerable patient population.

Study Procedures Recruitment and Data Collection: Eligible families seen in the Pediatric NF Clinic at VCU will be invited to participate via telephone or in person (depending on timing of clinic visit). Interested patients and parents/caregivers will provide informed consent, parental permission, and assent prior to data collection. Consented participants will be randomly allocated to the intervention (n=25) or control (n=25) groups via a computerized randomization program.

Data collection will occur at four timepoints: baseline (T0), 3-months (T1), 6-months (T2), and 7-months (T3). At T0 through T2, patients will complete standardized assessment batteries for neurocognitive functioning; and, patients, parents, and teachers will complete standardized questionnaires. All measures used within the present study are well validated and can be administered longitudinally within these time intervals with acceptable test-retest reliability. At T3, families in the intervention group will complete semi-structured qualitative interviews about the feasibility, acceptability, and desirability of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible if they are English-speaking children and adolescents between the ages of 6 to 16 years diagnosed with NF who are currently followed by the Pediatric NF Clinic at VCU. Patients are eligible if they currently have a diagnosis of ADHD or do not have a diagnosis of ADHD.
* At least one parent/caregiver must be actively involved in the patient's care and able to complete study-related questionnaires at baseline, 3-, and 6-months; and the exit interview at 7-months. Parents are eligible if they if they are English-speaking adults 18+ years old and self-identify as the parent or guardian of the patient.

Exclusion Criteria:

* Presence of serious, chronic comorbid condition (asthma and ADHD are not exclusionary criteria), presence of serious cognitive/learning impairment (e.g., down syndrome, moderate to severe intellectual disability or developmental disability), temporary foster care or residential care placement with no known plans to remain with foster parent for at least one year, presence of serious ongoing psychiatric disorder that prevents patient or family member from accurately completing questionnaires, and/or family anticipates moving in the next 12 months.
* No subject will be excluded on the basis of gender or ethnicity.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change in intellectual function | Baseline, 3 months, 6 months
  Intellectual function will be assessed using the Wechsler Intelligence Scale for Children (WISC) adapted to the age of the child. The child is asked to perform a variety of intellectual tasks. Overall and subscale scores are calculated by summing the number of correct answers. Higher scores indicate better intellectual function.
Change in neurocognitive function | Baseline, 3 months, 6 months
  Neurocognitive function will be assessed using the NIH Toolbox Cognitive Test Battery (NCTB). The NCTB is a standardized set of brief measures. Tasks are completed on a tablet and scores can be evaluated separately or as composite scores. Scores are normalized with a score of 100 being average, lower scores indicating lower neurocognitive function, and higher scores indicating higher cognitive function.

SECONDARY OUTCOMES:
Satisfaction with intervention | 7 months
  Quantitative: Feasibility exit interview

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Rohan, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No